CLINICAL TRIAL: NCT04291313
Title: Vitamin D Deficiency in Pregnancy - Identifying Associations and Mechanisms Linking Maternal Vitamin D Deficiency to Placental Dysfunction and Adverse Pregnancy Outcomes
Brief Title: Vitamin D in Pregnancy
Acronym: GRAVITD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GRAVITD
Record Dates: First submitted 2020-02-17; First posted 2020-03-02 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Vitamin D Deficiency; Pre-Eclampsia; Fetal Growth Retardation; Gestational Diabetes
MeSH Terms: conditions — Vitamin D Deficiency; Pre-Eclampsia; Fetal Growth Retardation; Diabetes, Gestational | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Treatment is blinded for participants and for the caretakers including nurses, midwifes and obstetricians.
  The investigators do not participate in diagnosing patients and are not blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Current recommended dose of vitamin D (Placebo Comparator): Women in this study arm receive 10 µg of vitamin D3 per day, which is the dose in a standard prenatal multivitamin and the dose currently recommended by the Danish Health Authorities to all pregnant women. They will receive a prenatal vitamin containing 10µg of vitamin D + a placebo supplement.
  Interventions: Dietary Supplement: Vitamin D3 (10µg)
- Higher dose of vitamin D (Experimental): Women in this arm receive 90µg of vitamin D3 per day: 10 µg from a standard prenatal multivitamin + an additional supplement containing 80µg of vitamin D3.
  Interventions: Dietary Supplement: Vitamin D3 (90µg)

INTERVENTIONS:
Dietary Supplement: Vitamin D3 (90µg) — The intervention is a higher dose of vitamin D than what is currently recommended to Danish pregnant women
  Arms: Higher dose of vitamin D
Dietary Supplement: Vitamin D3 (10µg) — This intervention serves as a control as they get the current recommended vitamin D dose
  Arms: Current recommended dose of vitamin D

SUMMARY:
Danish pregnant women are recommended ad daily vitamin D supplement of 10 µg. Despite the fact that 9 out of 10 women take vitamin D supplements, more than 40% of pregnant women are vitamin D deficient, putting them at an increased risk of pregnancy complications like fetal growth restriction and pre-eclampsia. Our hypothesis is that pregnant women would benefit from an increased intake og vitamin D and that an intake of 90µg/day can reduce the prevalence of placenta-related pregnancy complications. Combining a double-blinded randomized trial (10µg vs.90µg) with collection of placental material, we want to test if the prevalence of pregnancy complications is reduced and explore how vitamin D affects placenta to improve our understanding of the disease pathology and risk factors.

DETAILED DESCRIPTION:
As vitamin D (vit-D) is essential for growth and linked to placental function, health authorities recommend a daily 10µg vit-D supplement in pregnancy. Despite the fact that 9 out of 10 women take supplements, more than 40% of pregnant women are vit-D deficient, putting them at an increased risk of pregnancy complications like fetal growth restriction and pre-eclampsia. These conditions affect 6-10 % of all pregnancies, increasing the risk of preterm delivery, perinatal morbidity and mortality. In worse case, preeclampsia may also be fatal for the pregnant women herself. Around 20% of vit-D intake comes from the diet (e.g. fish, egg yolk) and the rest from sun-exposure. However, in Denmark, there is not enough sunlight from October to March to fuel vit-D synthesis underlining the need for supplementation. The high prevalence of vit-D deficiency indicates that current guidelines are not sufficient. Indeed, today´s recommendations date back to a small-scale 1986 Norwegian study not taking into account dietary differences such as the high intake of fish in Norway. Since then, accumulating evidence has linked exposure to pregnancy complications and vit-D deficiency per see to long-term health problems in the affected children. This include a higher risk of asthma, cardiovascular disease, diabetes, obesity schizophrenia, neurodevelopmental problems and multiple sclerosis. Notably, the affected women also suffer an increased risk of disease, e.g. heart disease in later life. Vitamin D supplements in the range of 90-100 µg are safe in pregnancy, but it is not yet known if and to what extent increased vitamin D supplementation prevents pregnancy-related diseases. Combining clinical testing of 90 µg vitamin D supplements, with identification of which placental pathways that are affected by vit-D would considerably improve our understanding of disease pathophysiology and the role of vit-D and improve the health of future generations in an easily implementable way.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women attending the nuchal translucency scan in week 11-13 of gestation as part of the national prenatal screening program

Exclusion Criteria:

* Age< 18 years
* Women with calcium metabolism disorders,
* Women who gets doctor prescribed vitamin D treatment
* Women with chronic kidney disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2020-06-08 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
The prevalence of pre-eclampsia (PE) | From 20 weeks of gestation to delivery
  The effect of 90 μg on the prevalence of PE
The prevalence of fetal growth retardation (FGR) | From 20 weeks of gestation to delivery
  The effect of 90 μg on the prevalence of FGR
The prevalence of gestational diabetes (GDM) | From 20 weeks of gestation to delivery
  The effect of 90 μg on the prevalence of GDM

SECONDARY OUTCOMES:
Changes in the placental expression of genes- and proteins related to vitamin D, evaluated using Next Generation Sequencing (NGS), quantitative Polymerase Chain Reaction (qPCR), methylation (Bisulfite conversion) and western blotting. | At delivery
  Characterization of the changes in the placenta as a result of vitamin D deficiency in healthy women including evaluation of the effect of BMI on placental function and vitamin D metabolism.
  NGS will be used to obtain a pathway analysis of differences between groups. Important findings from NGS will be verified on genetic and protein levels by qPCR and Western blotting respectively. Findings from NGS, qPCR and western blotting will be combined to characterize the changes in placentas from vitamin D deficient women compared to vitamin D sufficient women stratified by BMI.
  Further, changes in the expression of pivotal genes/proteins related to vitamin D metabolism (CYP2R1, CYP27B1, CYP24A1, Vitamin D receptor) will be investigated using qPCR, methylation analysis and western blotting. Findings from qPCR (gene level) methylation (gene level) and western blotting (protein level) are combined to characterize changes in placentas.
  Analyses will be done in subgroups of participants
Changes in the placental expression of genes- and proteins related to vitamin D and the pathogenesis of PE, FGR and GDM in placental tissue from complicated pregnancies compared to uncomplicated pregnancies, evaluated using NGS, qPCR and western blotting | At delivery
  Identification of changes in placental expression of genes and proteins related to the pathogenesis of PE, FGR and GDM and their relationship to vitamin D sensitive placental functions in complicated pregnancies (PE, FGR, GDM) compared to healthy uncomplicated pregnancies.
  NGS will be used to obtain a pathway analysis of differences in the gene expression between complicated pregnancies (PE, FGR, GDM) and healthy uncomplicated pregnancies. Important findings from the NGS studies will be verified on genetic and protein levels by qPCR and Western blotting. Findings from the NGS and the verifying results from qPCR (gene level) and western blotting (protein level) will be combined to characterize the changes in placentas from complicated pregnancies (PE, FGR, GDM) compared to healthy uncomplicated pregnancies.
  Analyses will be done in subgroups of participants
Birthweight | At delivery
  The effect of 90 μg vitamin D on birthweight.
Size related to gestational age | At delivery
  The effect of 90 μg vitamin D on size related to gestational age (Small for Gestational Age;SGA, Appropriate for Gestational Age; AGA, Large for Gestational Age;LGA)
The prevalence of preterm birth | At delivery
  The effect of 90 μg vitamin D on the prevalence of preterm birth (birth < 37 weeks of gestation).
The prevalence of postterm birth | At delivery
  The effect of 90 μg vitamin D on the prevalence of postterm birth (birth > 40 weeks of gestation)
The prevalence of gestational hypertension | From 20 weeks of gestation to delivery
  The effect of 90 μg vitamin D on the prevalence of gestational hypertension (>140/90)
Mode of delivery | At delivery
  Mode of delivery
The prevalence of infection during delivery | At delivery
  Infection during delivery (incl. use of antibiotics)
Admission to the neonatal ward | The first two weeks after birth
  Admission of the new born child to the neonatal ward
Prevalence of post partum hemorrhage > 500 ml | The first 24 hours after delivery
  The effect of 90 μg vitamin D on the prevalence of post partum hemorrhage > 500 ml

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Department of Biomedicine, University of Aarhus, Aarhus
  - Randers Regional Hospital, Randers

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vestergaard AL, Christensen M, Andreasen MF, Larsen A, Bor P. Vitamin D in pregnancy (GRAVITD) - a randomised controlled trial identifying associations and mechanisms linking maternal Vitamin D deficiency to placental dysfunction and adverse pregnancy outcomes - study protocol. BMC Pregnancy Childbirth. 2023 Mar 15;23(1):177. doi: 10.1186/s12884-023-05484-x. PMID 36922777